CLINICAL TRIAL: NCT04527328
Title: A Randomized, Double-Blind, Phase 2a Study to Evaluate the Tolerability, Feasibility, and Efficacy of AKST1210 in Patients on Hemodialysis With Cognitive Impairment Associated With End-Stage Renal Disease
Brief Title: A Study to Assess the Tolerability and Efficacy of AKST1210 in Patients on Hemodialysis With Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alkahest, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AKST1210-201
Record Dates: First submitted 2020-05-22; First posted 2020-08-26 (Actual); Results first posted 2022-12-12 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-11

CONDITIONS: Cognitive Impairment; End Stage Renal Disease
Keywords: Renal disease; Renal failure, chronic; End stage kidney disease; Chronic kidney failure; Kidney disease; Cognitive decline; Mental deterioration; Cognition disorder
MeSH Terms: conditions — Cognitive Dysfunction; Kidney Failure, Chronic; Kidney Diseases; Cognition Disorders | interventions — Renal Dialysis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- AKST1210 (Experimental): The AKST1210 column will be connected to the dialysis circuit during each dialysis session.
  Interventions: Device: AKST1210; Procedure: Hemodialysis
- Sham Control (No Intervention) (Sham Comparator): A covered surrogate object of similar size and shape as the investigational device
  Interventions: Other: Sham Control (No Intervention); Procedure: Hemodialysis

INTERVENTIONS:
Device: AKST1210 — AKST1210
  Arms: AKST1210
Other: Sham Control (No Intervention) — A covered surrogate object of similar size and shape as the investigational device
  Arms: Sham Control (No Intervention)
Procedure: Hemodialysis — Hemodialysis

SUMMARY:
This study will evaluate the tolerability, feasibility, and efficacy of the AKST1210 column in subjects with end-stage renal disease with cognitive impairment (ESRD-CI) undergoing hemodialysis 3 times per week.

DETAILED DESCRIPTION:
In this study, approximately 26 men and women on dialysis due to end stage renal disease and who have cognitive impairment will be randomly assigned to receive AKST1210 or control during each hemodialysis session for 3 months. The primary objective is to assess the safety and tolerability of AKST1210, and secondary objectives include changes in cognitive assessments as well as the feasibility of using AKST1210 in this setting.

ELIGIBILITY:
Inclusion Criteria:

* On chronic hemodialysis due to end-stage renal disease for ≥ 12 months.
* Score on the Montreal Cognitive Assessment (MoCA) ≥ 16 and ≤ 23.
* Body mass index (BMI) ≥ 20 and ≤ 36.
* The subject must be able to follow the study protocol, receive the treatment in the established timeframe, and continue during the follow-up interval.
* The subject must have sufficient visual and auditory acuity to reliably complete all study assessments.
* Provided a signed and dated informed consent form.

Exclusion Criteria:

* Subjects for whom adequate anticoagulation cannot be achieved. Use of antiplatelet drugs (e.g., aspirin or clopidogrel) is allowed.
* History of hypersensitivity to heparin.
* Pregnant or breast-feeding women or women who are planning to become pregnant.
* Clinically significant abnormalities on Screening ECG including QT interval corrected for heart rate (QTc) (using Fridericia's correction formula) of ≥ 500 ms in men and ≥ 520 ms in women.
* Clinically significant and unexpected abnormalities in this patient population in complete blood count, complete metabolic panel, coagulation, and thyroid stimulating hormone (TSH).
* Subjects with a hemoglobin level < 9.0 g/dL.
* Concurrent or recent participation in another investigational clinical trial. Prior clinical trial subjects must have discontinued investigational agents at least 30 days prior to Screening.
* Subjects planning to receive renal transplantation during the study.
* Any other condition and/or situation that the investigator believes may interfere with the safety of the subject, study conduct, or interpretation of study data.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-04-28 (Actual); Primary Completion 2021-06-04 (Actual); Study Completion 2021-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alkahest Medical Monitor, Study Director — Alkahest, Inc.
Locations (4):
- United States (4):
  - Renal Consultants Medical Group, Granada Hills, California
  - Valley Renal Medical Group, Northridge, California
  - Orlando Clinical Research Center, Orlando, Florida
  - US Renal Care Kidney Research, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- AKST1210: The AKST1210 column will be connected to the dialysis circuit during each dialysis session.
  AKST1210: AKST1210 column
  Hemodialysis: Hemodialysis
Period: Overall Study
Arm/Group | AKST1210 | Sham Control (No Intervention)
Started | 5 | 5
AKST1210 S-15 or Control | 5 | 5
AKST1210 S-25 or Control | 5 | 5
AKST1210 S-35 or Control | 4 | 5
Completed (Subjects who completed the End of Study (follow-up) visit) | 3 | 5
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- AKST1210 Device: The AKST1210 column will be connected to the dialysis circuit during each dialysis session.
  AKST1210: AKST1210 column
  Hemodialysis: Hemodialysis
- Total: Total of all reporting groups
Arm/Group | AKST1210 Device | Sham Control (No Intervention) | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (10.78) | 61.6 (10.6) | 61 (10.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 4 | 5 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 2 | 3 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events Assessed by Intensity
Description: Number of participants with Treatment-Emergent Adverse Events (TEAE) assessed by Intensity (mild, moderate, or severe) coded by the Medical Dictionary for Regulatory Activities (MedDRA)
Time Frame: Baseline to Week 14
Measure: Number; unit: participants
Arm/Group | AKST1210 | Sham Control (No Intervention)
Number analyzed (Participants) | 5 | 5
participants
  Mild TEAE | 0 | 1
  Moderate TEAE | 2 | 2
  Severe TEAE | 2 | 0

2. Secondary Outcome: Tolerability as Measured by the Number of Subjects Who Complete Each Treatment Period
Description: The number of subjects will be summarized by AKST1210 column size (small, S-15; medium, S-25; and large, S-35) and control for subjects who completed all visits in the treatment period
Time Frame: Baseline to Week 12
Measure: Number; unit: participants
Groups:
- AKST1210 (S-15): Extracorporeal device (S-15, 150 mL capacity) for use in conjunction with dialysis
- AKST1210 (S-25): Extracorporeal device (S-25, 250 mL capacity) for use in conjunction with dialysis
- AKST1210 (S-35): Extracorporeal device (S-35, 350 mL capacity) for use in conjunction with dialysis
- Control Column: A sham control with no effect on the dialyzed blood will be used to mimic the appearance of an in-line AKST1210 device
Arm/Group | AKST1210 (S-15) | AKST1210 (S-25) | AKST1210 (S-35) | Control Column
Number analyzed (Participants) | 5 | 5 | 4 | 5
participants | 5 | 5 | 3 | 5

3. Secondary Outcome: Number of Participants Who Discontinued Due to Intradialytic Hypotension (IDH)
Description: The number and percentage of subjects requiring early discontinuation from study treatment due to IDH summarized by treatment group
Time Frame: Baseline to Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | AKST1210 | Sham Control (No Intervention)
Number analyzed (Participants) | 5 | 5
Participants | 1 | 0

4. Secondary Outcome: Change From Baseline in Montreal Cognitive Assessment (MoCA)
Description: Change from baseline to EOS in the total Montreal Cognitive Assessment (MoCA) score, which assesses executive functions, naming, attention and concentration, language, abstraction, delayed recall, and orientation. The MoCA has a total score from 0 to 30 whereby all sub sections are summed. The scoring breakdown for all sub sections includes the following: Visuospatial and executive functioning: 0-5 points, naming: 0-3 points, attention: 0-6 points, language: 0-3 points, abstraction: 0-2 points, delayed recall: 0- 5 points, orientation: 0-6 points. 1 point is added to the test-taker's score if they have 12 years or less of formal education. Higher scores in all sub categories and total score indicate better cognition. The Mean change from baseline is the post-treatment value minus baseline value.
Time Frame: Screening to Week 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AKST1210 | Sham Control (No Intervention)
Number analyzed (Participants) | 2 | 5
score on a scale
  Total Score | 1.0 (1.41) | 0.6 (1.14)
  Visuospatial / Executive | 0.5 (0.71) | -0.2 (1.30)
  Naming | 0.5 (0.71) | 0.0 (0.00)
  Attention | -1.0 (0.00) | 0.2 (0.45)
  Language | 0.0 (0.00) | 0.2 (0.84)
  Abstraction | 0.5 (0.71) | 0.0 (1.00)
  Delayed Recall | 2.0 (0.00) | 0.4 (1.52)
  Orientation | 0.0 (0.00) | -0.2 (0.45)

5. Secondary Outcome: Change From Baseline in Computer-based Cognitive Assessment (CogState) Composite Score
Description: Mean change from baseline to End of Treatment in CogState test battery composite scores. The CogState test battery is a simple, brief computerized battery designed to assess cognitive function in several areas including verbal learning, psychomotor function, visual attention, working memory, executive function, and verbal delayed recall. Higher scores indicate better outcomes for all composite scores. All composite scores have a range of -16 to 10. Z-Scores between ≥ 1 and < 1.5 standard deviations (SD) below age-matched normative data are considered minor cognitive impairment. Z-Scores between ≥ 1.5 and < 2 SD below age-matched normative data are considered mild cognitive impairment. Z-Scores ≥ 2 SD below age matched normative data are considered major cognitive impairment consistent with dementia.
Time Frame: Baseline to Week 12
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | AKST1210 | Sham Control (No Intervention)
Number analyzed (Participants) | 4 | 5
Z-score
  Global Composite Score | -0.1 (2.07) | 0.4 (0.84)
  Episodic Memory Domain Composite Score | -0.2 (1.30) | 0.5 (0.37)
  Attention Domain Composite Score | 0.0 (3.86) | 0.6 (2.12)
  Executive Function Domain Composite Score | 0.0 (1.70) | 0.1 (0.58)
  Psychomotor Function Composite Score | 0.6 (3.80) | 0.7 (2.53)
  Working Memory Composite Score | -0.3 (2.74) | 0.6 (1.82)
  Verbal Learning Composite Score | -0.1 (1.71) | 0.3 (0.57)

6. Secondary Outcome: Change From Baseline in Quality of Life Per the Short-Form Health Survey (SF-36)
Description: Mean change from baseline in quality of life per the Short-Form Health Survey (SF-36), which evaluates quality of life measures. All scores range from 0 to 100 with higher scores indicating less disability. An increase or decrease in the mental health summary score or physical health summary score from baseline indicates a more favorable health status or a more unfavorable health status, respectfully, in the subject's quality of life related to mental or physical health.
Time Frame: Baseline to Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AKST1210 | Sham Control (No Intervention)
Number analyzed (Participants) | 4 | 5
score on a scale
  Physical Health Score | -9.6 (12.35) | -3.4 (9.66)
  Mental Health Score | 0.7 (6.59) | 4.1 (9.71)

7. Secondary Outcome: Change From Baseline in the Patient Health Questionnaire-9 (PHQ-9)
Description: Change from baseline to EOS in the Patient Health Questionnaire-9 (PHQ-9), which evaluates the severity of depression. Symptoms are rated from 0 (not at all) to 3 (nearly every day) and scores are summated for each subject across the 9 items. The total score range is 0-27. An increase or decrease in the PHQ-9 total score from baseline indicates greater severity or less severity, respectfully, in the subject's state of depression.
Time Frame: Baseline to Week 14
Population: Number analyzed for each row title reflects available data. Subjects with missing data at the End of Study visit are excluded.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AKST1210 | Sham Control (No Intervention)
Number analyzed (Participants) | 4 | 5
score on a scale | 3.5 (5.20) | -1.2 (1.92)

8. Secondary Outcome: Change From Baseline in Sleep Quality Per the Pittsburgh Sleep Quality Index (PSQI)
Description: Change from baseline in sleep quality as measured by the Sleep Quality Per the Pittsburgh Sleep Quality Index (PSQI), which measures the quality and patterns of sleep in older adults. It differentiates "poor" from "good" sleep by measuring 7 domains: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction over the last month. The subject self-rates each of these 7 areas of sleep. The score for each domain ranges from 0 to 3, whereby higher scores for each reflect the negative (worse) extreme on the Likert Scale. The sum of all 7 domains is used to compute the total score (0 to 21). A global sum of "5" or greater indicates a "poor" sleeper. An increase or decrease in the PSQI total score from baseline indicates worsening or improvement, respectfully, in the subject's overall sleep quality.
Time Frame: Baseline to Week 12
Population: Number analyzed for each row title reflects available data. Subjects with missing data at the End of Treatment visit are excluded.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AKST1210 | Sham Control (No Intervention)
Number analyzed (Participants) | 4 | 5
score on a scale
  Total Score: number analyzed (Participants) | 3 | 4
  Total Score | 0.0 (4.58) | 0.8 (2.22)
  Sleep Quality: number analyzed (Participants) | 3 | 5
  Sleep Quality | 0.3 (0.58) | 0.2 (0.45)
  Sleep Latency: number analyzed (Participants) | 3 | 5
  Sleep Latency | -0.3 (1.53) | 0.2 (0.84)
  Sleep Duration | -0.3 (0.50) | 0.0 (0.71)
  Habitual Sleep Efficiency | 0.0 (1.63) | 0.6 (1.34)
  Sleep Disturbances: number analyzed (Participants) | 3 | 4
  Sleep Disturbances | 0.0 (0.00) | 0.0 (0.00)
  Use of Sleep Medication: number analyzed (Participants) | 3 | 5
  Use of Sleep Medication | 0.0 (0.0) | 0.0 (0.0)
  Daytime Dysfunction over the Last Month: number analyzed (Participants) | 3 | 4
  Daytime Dysfunction over the Last Month | 0.3 (0.58) | 0.5 (0.58)

9. Secondary Outcome: Change From Baseline in Fatigue Per the Fatigue Questionnaire - Functional Assessments of Chronic Illness Therapy (FACIT)
Description: Change from baseline to End of Treatment in fatigue as measured by the Functional Assessments of Chronic Illness Therapy (FACIT), which measures an individual's level of fatigue during their usual daily activities over the past week. The level of fatigue for each question is measured on a 4-point Likert scale (4 = not at all fatigued to 0 = very much fatigued). The total score range is 0 to 52. To get this total, each question answered is scored individually, summed, multiplied by 13, and lastly divided by the number of questions answered. The higher the total score, the better the quality of life.
Time Frame: Baseline to Week 12
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AKST1210 | Sham Control (No Intervention)
Number analyzed (Participants) | 4 | 5
score on a scale | -0.5 (10.12) | 0.2 (5.17)

10. Secondary Outcome: Number of Participants Who Discontinued Due to Anemia.
Description: The number and percentage of subjects with any anemia leading to discontinuation from AKST1210/control will be summarized by treatment group and total.
Time Frame: Baseline to Week 12
Measure: Count of Participants; unit: Participants
Arm/Group | AKST1210 | Sham Control (No Intervention)
Number analyzed (Participants) | 5 | 5
Participants | 0 | 0

11. Secondary Outcome: Tolerability as Measured by the Percentage of Subjects Who Complete Each Treatment Period
Description: The percentage of subjects will be summarized by AKST1210 column size (small, S-15; medium, S-25; and large, S-35) and control for subjects who completed all visits in the treatment period
Time Frame: Baseline to Week 12
Measure: Number; unit: percentage of participants
Groups:
- AKST1210 (S-15): The AKST1210 (S-15, 150 mL) column will be connected to the dialysis circuit during each dialysis session.
- AKST1210 (S-25): The AKST1210 (S-25, 250 mL) column will be connected to the dialysis circuit during each dialysis session.
- AKST1210 (S-35): The AKST1210 (S-35, 350 mL) column will be connected to the dialysis circuit during each dialysis session.
Arm/Group | AKST1210 (S-15) | AKST1210 (S-25) | AKST1210 (S-35) | Control Column
Number analyzed (Participants) | 5 | 5 | 4 | 5
percentage of participants | 100.00 | 100.00 | 75.00 | 100.00

12. Secondary Outcome: Tolerability as Measured by the Number of Subjects Who Complete the Run-In Period.
Description: The number of subjects who completed the run-in period prior to randomization and initiation of study treatment. Subjects who met all eligibility criteria assessed during screening were monitored during a two-week run-in period for ongoing assessment of eligibility, safety, and baseline assessments prior to randomization and initiation of study treatment.
Time Frame: Week -2 (Day -14) to Week -1 (Day -1)
Measure: Number; unit: participants
Groups:
- Participants Who Entered Run-in: The total number of participants who entered into the run-in period
Arm/Group | Participants Who Entered Run-in
Number analyzed (Participants) | 11
participants | 10

13. Secondary Outcome: Tolerability as Measured by the Percentage of Subjects Who Complete the Run-in Period
Description: The percentage of subjects who completed the run-in period prior to randomization and initiation of study treatment. Subjects who met all eligibility criteria assessed during screening were monitored during a two-week run-in period for ongoing assessment of eligibility, safety, and baseline assessments prior to randomization and initiation of study treatment.
Time Frame: Week -2 (Day -14) to Week -1 (Day -1)
Measure: Number; unit: percentage of participants
Arm/Group | Participants Who Entered Run-in
Number analyzed (Participants) | 11
percentage of participants | 90.9

14. Secondary Outcome: Tolerability as Measured by the Number of Subjects Who Completed All Visits.
Description: The number of subjects will be summarized by column size (small, S-15; medium, S-25; and large, S-35) and control for subjects who completed all visits
Time Frame: Baseline to Week 14
Population: One subject completed all visits in the S-25 treatment period but discontinued prior entering the S-35 treatment period. Another subject completed all visits in the S-35 treatment period but discontinued prior completing the End of Study Follow-up visit
Measure: Number; unit: participants
Arm/Group | AKST1210 (S-15) | AKST1210 (S-25) | AKST1210 (S-35) | Control Column
Number analyzed (Participants) | 5 | 5 | 4 | 5
participants | 5 | 5 | 3 | 5

15. Secondary Outcome: Tolerability as Measured by the Percentage of Subjects Who Completed All Visits.
Description: The percentage of subjects will be summarized by column size (small, S-15; medium, S-25; and large, S-35) and control for subjects who completed all visits
Time Frame: Baseline to Week 14
Population: Of the 4 subjects entering into Treatment Period 3 (S-35), one subject did not complete the End of Study follow-up visit
Measure: Number; unit: percentage of participants
Arm/Group | AKST1210 (S-15) | AKST1210 (S-25) | AKST1210 (S-35) | Control Column
Number analyzed (Participants) | 5 | 5 | 4 | 5
percentage of participants | 100.00 | 100.00 | 75.00 | 100.00

ADVERSE EVENTS:
Time Frame: Approximately 16-20 weeks (up to 4 weeks for screening and 14 weeks on study, inclusive of the 2-week run-in period)
Description: AEs were captured beginning at time of informed consent through EOS. AE status was followed by the investigator until resolved or considered stable, unless the subject was lost to follow up. Reporting of TEAEs and AEs followed the pre-specified analyses per the Statistical Analysis Plan (SAP) in which total safety events were summarized by randomization arm (AKST1210 combined or Control combined).
Arm/Group | AKST1210 | Sham Control (No Intervention)
All-Cause Mortality (participants affected / at risk) | 1/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 2/5 | 0/5
Other Adverse Events (participants affected / at risk) | 3/5 | 3/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AKST1210 (N=5) | Sham Control (No Intervention) (N=5)
Cardiac arrest (Cardiac disorders) | 1 | 0
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AKST1210 (N=5) | Sham Control (No Intervention) (N=5)
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 0 | 1
Lipase increased (Investigations) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Dialysis hypotension (Vascular disorders) | 2 | 0
Hypotension (Vascular disorders) | 1 | 1

LIMITATIONS AND CAVEATS:
After the study was closed, unreliable data was identified at a single study site and has not been presented here.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2020-02-14): https://cdn.clinicaltrials.gov/large-docs/28/NCT04527328/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-25): https://cdn.clinicaltrials.gov/large-docs/28/NCT04527328/SAP_001.pdf